CLINICAL TRIAL: NCT01662427
Title: Nocturnal Parkinson's Disease Symptoms Study Group
Status: Completed | Type: Observational
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Roongroj Bhidayasiri, Associate Professor, Chulalongkorn University
Other Study IDs: 6222012
Record Dates: First submitted 2012-08-07; First posted 2012-08-10 (Estimated); Last update posted 2013-08-20 (Estimated); Status verified 2013-08

CONDITIONS: Parkinson's Disease
Keywords: Quality of life; Noctural Parkinson's Disease Symptoms
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Questionniare
  Interventions: Other: Questionaire to assess Noctural Parkinson's Disease Symptoms

INTERVENTIONS:
Other: Questionaire to assess Noctural Parkinson's Disease Symptoms — Questionaire to assess Noctural Parkinson's Disease Symptoms and quality of life

SUMMARY:
To study associate factor of Noctural Parkinson's Disease Symptoms and quality of life in Parkinson's disease patients and caregivers.

ELIGIBILITY:
Inclusion Criteria:

Idiopathic Parkinson's disease patient

Exclusion Criteria:

1. Patient with Secondary Parkinsonism eg.Drug-induced Parkinsonism, Vascular Parkinsonism, exposure to toxin, Encephalitis
2. Patient with Atypical Parkinsonial Syndromes eg. Parkinson-plus syndrome, Progressive Supranuclear Palsy (PSP), Corticobasal Degeneration (CBD)
3. Patient with Heredodegenerative parkinsonism eg. Spinocerebellar ataxias, Wilson's disease, Juvenile Huntington's disease

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Parkinson's disease patient and care givers
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2012-11; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
To assess Noctural Parkinson's Disease Symptoms

SECONDARY OUTCOMES:
To assess quality of life in Parkinson's Disease patient
To assess quality of life in caregiver of Parkinson's Disease patient

CONTACTS AND LOCATIONS:
Locations (1):
- Roongroj Bhidayasiri, Pathumwan, Bangkok, Thailand